CLINICAL TRIAL: NCT02362724
Title: Evaluation of the CooperVision, Inc. Sapphire and Pearl Silicone Hydrogel Daily Wear Contact Lenses When Used for Frequent Replacement for Up to One (1) Month of Daily Wear.
Brief Title: Evaluation of Investigational (Frequent Replacement) FRP Lens for Daily Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FC131202
Record Dates: First submitted 2015-02-02; First posted 2015-02-13 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2015-12

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sapphire (Experimental): Subjects randomized to the experimental contact lens over the study duration
  Interventions: Device: Sapphire
- Pearl (Active Comparator): Subjects randomized to the active comparator contact lens over the study duration
  Interventions: Device: Pearl

INTERVENTIONS:
Device: Sapphire — silicone hydrogel contact lens
  Arms: Sapphire
Device: Pearl — silicone hydrogel contact lens
  Arms: Pearl

SUMMARY:
The purpose of the study is to compare the investigational contact lens to a marketed contact lens.

The study results were not used for design validation of investigational contact lens,

DETAILED DESCRIPTION:
The objective of this evaluation is to provide evidence supporting the claim that the performance of the Test Lens is substantially equivalent to that of the Control Lens when used in a one month (up to 30 days) recommended replacement, daily wear modality.

The study results were not used for design validation of investigational contact lens,

ELIGIBILITY:
Inclusion Criteria:

* Prior to being considered eligible to participate in this study, each subject MUST:

  1. Be at least 18 years of age as of the date of evaluation for the study.
  2. Have:

     1. Read the Informed Consent
     2. been given an explanation of the Informed Consent
     3. indicated understanding of the Informed Consent
     4. signed the Informed Consent document.
  3. Be willing and able to adhere to the instructions set forth in this protocol and able to keep all specified appointments.
  4. Be an adapted, current full-time silicone hydrogel or soft contact lens wearer. An adapted full-time wearer is defined as wearing contact lenses at least 5 days per week for at least 8 hours per day for at least one month prior to participation in the study.
  5. Possess or obtain prior to dispensing, wearable and visually functional (20/40 or better) eyeglasses.
  6. Be in good general health, based on his/her knowledge.
  7. Require spectacle lens powers between -0.50 and -8.00 diopters sphere with no more than 1.50 diopter of refractive astigmatism and be willing to wear contact lenses in both eyes.
  8. Have manifest refraction Snellen visual acuities (VA) equal to or better than 20/25 in each eye.
  9. To be eligible for lens dispensing, the subject must achieve 20/30 VA or better in each eye with the study lens and the investigator must judge the fit as acceptable or optimal.

Exclusion Criteria:

* Subjects may not be enrolled in this study if any of the following apply: The subject is currently or has:

  1. Wearing lenses in a monovision modality and is unwilling to be fit with distance lenses in both eyes for the duration of the study. NOTE: Subjects may not wear lenses in a monovision modality at any time during the study as it will interfere with the visual acuity analysis.
  2. Poor personal hygiene.
  3. Any active participation in another clinical trial during this trial or within 30 days prior to this study.
  4. To the best of the subject's knowledge, she is currently pregnant, is lactating or is planning a pregnancy within the next 3 months.
  5. A member, relative or household member of the investigator or of the investigational office staff.
  6. Has a known sensitivity to the ingredients used in the MPS approved for use in the study and is unable or unwilling to use the alternate care system.
  7. Previous refractive surgery; or current or previous orthokeratology treatment.
  8. Is aphakic or psuedophakic.
  9. Ocular or systemic disease such as, but not limited to: anterior uveitis or iritis (past or present), glaucoma, Sjögren's syndrome, lupus erythematosus, scleroderma, keratoconus or uncontrolled diabetes.
  10. The need for topical ocular medications or any systemic medication which might interfere with contact lens wear or require the lenses to be removed during the day.
  11. The presence of clinically significant (grade 2, 3 or 4) anterior segment abnormalities; or the presence of any inflammations such as iritis; or any infection of the eye, lids, or associated structures.
  12. A known history of corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates, iritis, bacterial or fungal infections.
  13. A history of papillary conjunctivitis that has interfered with contact lens wear.
  14. Slit lamp findings that would contraindicate contact lens wear, including but not limited to:

      * Pathological dry eye or associated dry eye symptoms with decreased tear levels and punctuate staining > Grade 2
      * Pterygium
      * Corneal scars within the visual axis
      * Neovascularization or ghost vessels > 1.0 mm in from the limbus
      * Giant papillary conjunctivitis (GPC) of > Grade 2
      * Anterior uveitis or iritis
      * Seborrheic eczema, seborrheic conjunctivitis or blepharitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Saltzman, MD, FACOG, Study Chair — Sterling IRB
Locations (6):
- United States (6):
  - Eric M White OD, Inc., San Diego, California
  - Office of Mark E Nakano, O.D., Torrance, California
  - Advanced Family Eye Care, Denver, North Carolina
  - Quinn Foster & Associates, Athens, Ohio
  - Primary Eyecare Group, P.C., Brentwood, Tennessee
  - Premier Vision Services, LLC, Amarillo, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Sapphire: Subjects were randomized in a 2:1(Test: Control) ratio to the experimental contact lens over the study duration
  Sapphire: silicone hydrogel contact lens
- Pearl: Subjects were randomized in a 2: 1 ratio (Test: Control) to the active comparator contact lens over the study duration
  Pearl: silicone hydrogel contact lens
Period: Overall Study
Arm/Group | Sapphire | Pearl
Started | 59 | 30
Completed | 53 | 29
Not Completed | 6 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sapphire | Pearl | Total
Number analyzed (Participants) | 59 | 30 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 30 | 89
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (8.820) | 33.3 (8.890) | 32.9 (8.800)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 18 | 58
  Male | 19 | 12 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  White | 47 | 23 | 70
  Japanese | 9 | 5 | 14
  Black | 1 | 1 | 2
  Hispanic | 1 | 1 | 2
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 59 | 30 | 89

OUTCOME MEASURES:

1. Primary Outcome: Slit Lamp Findings for Epithelial Edema
Description: Slit Lamp Findings for Epithelial Edema on a grade of 0-4 (0 NONE: No microcysts; normal transparency, 1 TRACE: 1 to 20 microcysts; barely discernible local epithelial haziness, 2 MILD: 21 to 50 microcysts; faint but definite localized or generalized haziness, 3 MODERATE: 51 to 100 microcysts; significant localized or generalized haziness, 4 SEVERE: >100 microcysts; definite widespread epithelial cloudiness giving a dull glass appearance to the cornea, or numerous coalescing bullae)
Time Frame: Baseline (After lens dispensing)
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 53 | 29
Number analyzed (Eyes) | 106 | 58
Eyes
  Grade 0 | 106 | 58
  Grade 1 | 0 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

2. Primary Outcome: Slit Lamp Findings for Epithelial Edema
Description: as for outcome 1
Time Frame: 1 Month
Population: Data for two test eyes and two control eyes were not collected.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 52 | 28
Number analyzed (Eyes) | 104 | 56
Eyes
  Grade 0 | 104 | 56
  Grade 1 | 0 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

3. Primary Outcome: Slit Lamp Findings for Stromal Edema
Description: Slit Lamp Findings for Stromal Edema on a grade of 0-4 (0 NONE: No edema, 1 TRACE: Just detectable clouding, 2 MILD: Faint corneal striae (2 or fewer), 3 MODERATE: Pronounced corneal striae (3), 4 SEVERE: Folds in Descemet's membrane and >4 pronounced striae)
Time Frame: Baseline (After lens dispensing)
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 53 | 29
Number analyzed (Eyes) | 106 | 58
Eyes
  Grade 0 | 106 | 58
  Grade 1 | 0 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

4. Primary Outcome: Slit Lamp Findings for Stromal Edema
Description: as for outcome 3
Time Frame: 1 month
Population: Data for two test eyes and two control eyes were not collected
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 52 | 28
Number analyzed (Eyes) | 104 | 56
Eyes
  Grade 0 | 104 | 56
  Grade 1 | 0 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

5. Primary Outcome: Slit Lamp Findings for Corneal Infiltrates
Description: Slit Lamp Findings for Corneal Infiltrates - Present, Absent
Time Frame: Baseline (After lens dispensing)
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 53 | 29
Number analyzed (Eyes) | 106 | 58
Eyes
  Present | 0 | 0
  Absent | 106 | 58

6. Primary Outcome: Slit Lamp Findings for Corneal Infiltrates
Description: Slit Lamp Findings for Corneal Infiltrates - Present, Absent
Time Frame: 1 Month
Population: Data for two test lens and two control lens were not collected
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 52 | 28
Number analyzed (Eyes) | 104 | 56
Eyes
  Present | 0 | 0
  Absent | 104 | 56

7. Primary Outcome: Slit Lamp Findings for Corneal Vascularization
Description: Slit Lamp Findings for Corneal Vascularization on a grade 0-4 (0 NONE: No vessel penetration, 1 TRACE: <1.00 mm vessel penetration, 2 MILD: >1.00 mm to <1.50 mm vessel penetration, 3 MODERATE: >1.50 mm to <2.00 mm vessel penetration, 4 SEVERE: Vessel penetration >2.00 mm)
Time Frame: Baseline (After lens dispensing)
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 53 | 29
Number analyzed (Eyes) | 106 | 58
Eyes
  Grade 0 | 103 | 52
  Grade 1 | 3 | 6
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

8. Primary Outcome: Slit Lamp Findings for Corneal Vascularization
Description: as for outcome 7
Time Frame: 1 month
Population: Data for two test eyes and two control eyes were not collected
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 52 | 28
Number analyzed (Eyes) | 104 | 56
Eyes
  Grade 0 | 101 | 52
  Grade 1 | 3 | 4
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

9. Primary Outcome: Slit Lamp Findings for Limbal Hyperemia
Description: Slit Lamp Findings for Limbal Hyperemia on a grade 0-4 (0 NONE: No hyperemia present, 1 TRACE: Slight regional hyperemia, 2 MILD: Diffuse hyperemia, 3 MODERATE: Marked regional or diffuse hyperemia, 4 SEVERE: Diffuse episcleral or scleral hyperemia)
Time Frame: Baseline (After lens dispensing)
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 53 | 29
Number analyzed (Eyes) | 106 | 58
Eyes
  Grade 0 | 77 | 48
  Grade 1 | 29 | 10
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

10. Primary Outcome: Slit Lamp Findings for Limbal Hyperemia
Description: as for outcome 9
Time Frame: 1 month
Population: Data for two test eyes and two control eyes were not collected.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 52 | 28
Number analyzed (Eyes) | 104 | 56
Eyes
  Grade 0 | 76 | 44
  Grade 1 | 28 | 12
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

11. Primary Outcome: Slit Lamp Findings for Bulbar Hyperemia
Description: Slit Lamp Findings for Bulbar Hyperemia on a grade 0-4 (0 NONE: No hyperemia present, 1 TRACE: Slight regional hyperemia, 2 MILD: Diffuse hyperemia, 3 MODERATE: Marked regional or diffuse hyperemia, 4 SEVERE: Diffuse episcleral or scleral hyperemia)
Time Frame: Baseline (After lens dispensing)
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 53 | 29
Number analyzed (Eyes) | 106 | 56
Eyes
  Grade 0 | 64 | 41
  Grade 1 | 42 | 17
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

12. Primary Outcome: Slit Lamp Findings for Bulbar Hyperemia
Description: as for outcome 11
Time Frame: 1 month
Population: Data for two test eyes and two control eyes were not collected.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 52 | 28
Number analyzed (Eyes) | 104 | 56
Eyes
  Grade 0 | 70 | 42
  Grade 1 | 33 | 14
  Grade 2 | 1 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

13. Primary Outcome: Slit Lamp Findings for Palpebral Conjunctiva
Description: Slit Lamp Findings for Palpebral Conjunctiva - Present, Absent
Time Frame: Baseline (After lens dispensing)
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 53 | 29
Number analyzed (Eyes) | 106 | 58
Eyes
  Present | 34 | 19
  Absent | 72 | 39

14. Primary Outcome: Slit Lamp Findings for Palpebral Conjunctiva
Description: Slit Lamp Findings for Palpebral Conjunctiva - Present, Absent
Time Frame: 1 month
Population: Data for two test eyes and two control eyes were not collected
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 52 | 28
Number analyzed (Eyes) | 104 | 56
Eyes
  Present | 47 | 20
  Absent | 57 | 36

15. Primary Outcome: Slit Lamp Findings for Other Findings
Description: Slit Lamp Findings for Other findings (conjunctival infection, corneal ulcers, iritis, lens adhesions and recurrent erosion) on a grade 0-4 (0 NONE, 1 TRACE, 2 MILD, 3 MODERATE, 4 SEVERE)
Time Frame: Baseline (After lens dispensing)
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 53 | 29
Number analyzed (Eyes) | 106 | 56
Eyes
  Grade 0 | 104 | 54
  Grade 1 | 2 | 4
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

16. Primary Outcome: Slit Lamp Findings for Other Findings
Description: as for outcome 15
Time Frame: 1 month
Population: Data for two test eyes and two control eyes were not collected
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Pearl
Number analyzed (Participants) | 52 | 28
Number analyzed (Eyes) | 104 | 56
Eyes
  Grade 0 | 101 | 54
  Grade 1 | 3 | 2
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Dispense up to one month on study lenses
Arm/Group | Sapphire | Pearl
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/30
Other Adverse Events (participants affected / at risk) | 7/59 | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sapphire (N=59) | Pearl (N=30)
Pappilary Conjuctivitis (Eye disorders) | 6 (6) | 1 (1)
Corneal Infiltrate (Eye disorders) | 0 (0) | 1 (1)
Foreign body Abrasion (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No